CLINICAL TRIAL: NCT01437072
Title: Changing Diabetes® World Tour a Study on the Association of Risk Factors and the Presence of Undiagnosed Diabetes in the Middle East, Northern Africa and Europe
Brief Title: Changing Diabetes® World Tour
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3934; U1111-1123-4683 (Other: WHO)
Record Dates: First submitted 2011-09-08; First posted 2011-09-20 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total study population
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — The screening test includes a combination of a risk assessment questionnaire and biochemical tests.

SUMMARY:
This study is conducted in the Middle East, Northern Africa and Europe. The aim of this study is to contribute to the design of a simple screening strategy for countries in scope, by exploring the association between risk factors and undiagnosed diabetes in a screening study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained

Exclusion Criteria:

* Subjects with known diabetes (exception: women with a history of gestational diabetes should not be excluded)
* Pregnant women or women who have given birth within less than a month
* Subjects suffering from severe illness
* Subjects with the inability to read and understand the information given (either due to illiteracy or vision problems) and therefore unable to give an informed consent
* Subjects with mental impairment
* Subjects treated with systemic cortico-steroids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Changing Diabetes® World Tour is designed as a mobile screening clinic staying for a minimum of 14 days in each location such as malls, public squares, etc. Subjects included in the study are either actively seeking to be screened, or are invited by subjects in their network already included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 8304 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
HbA1c (Glycosylated Haemoglobin) level | measured at the screening visit (only 1 visit during the 2 weeks stay of the bus in each country)

SECONDARY OUTCOMES:
Number of subjects with diabetes (type 1 and 2) | measured at the screening visit (only 1 visit during the 2 weeks stay of the bus in each country)
The presence of retinopathy | measured at the screening visit (only 1 visit during the 2 weeks stay of the bus in each country)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (3):
- Novo Nordisk Investigational Site, Paço de Arcos, Portugal
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia
- Novo Nordisk Investigational Site, Dubai, United Arab Emirates

REFERENCES:
- [Result] Handlos LN, Witte DR, Almdal TP, Nielsen LB, Badawi SE, Sheikh AR, Belhadj M, Nadir D, Zinai S, Vistisen D. Risk scores for diabetes and impaired glycaemia in the Middle East and North Africa. Diabet Med. 2013 Apr;30(4):443-51. doi: 10.1111/dme.12118. PMID 23331167
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com